CLINICAL TRIAL: NCT02809105
Title: Phase 3 Study of ASP0456 - A Double-blind, Placebo-controlled, Parallel-group, Comparative Study and an Open-label, Uncontrolled, Long-term Dosing Study in Patients With Chronic Constipation (Not Including Constipation Due to Organic Diseases) -
Brief Title: A Study of Oral Dosing of ASP0456 in Patients With Chronic Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0456-CL-1031
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Chronic Constipation
Keywords: Chronic constipation; Linaclotide; ASP0456
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part I ASP0456 (Experimental): ASP0456 will be administered orally for 4 weeks.
  Interventions: Drug: linaclotide
- Part I Placebo (Placebo Comparator): Placebo will be administered orally for 4 weeks.
  Interventions: Drug: Placebo
- Part II ASP0456 (Experimental): ASP0456 will be administered orally.
  Interventions: Drug: linaclotide

INTERVENTIONS:
Drug: linaclotide — Oral administration once daily
  Other Names: ASP0456
  Arms: Part I ASP0456; Part II ASP0456
Drug: Placebo — Oral administration once daily
  Arms: Part I Placebo

SUMMARY:
The objective of this study is to verify the efficacy and investigate the safety of the study drug when ASP0456 is administered orally for 4 weeks and 52 weeks.

DETAILED DESCRIPTION:
This study consists of two parts. In Part I, ASP0456 or placebo will be administered orally in a blind manner. In Part II, the long-term safety and efficacy of ASP0456 will be evaluated in patients who have participated in the study and completed the Part I.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SBM frequency for < 3 times/week, since ≥ 6 months prior to preliminary enrollment
* Patients with one or more related symptoms for ≥ 6 months prior to preliminary enrollment
* Patients at whom loose (mushy) or watery stools are rarely present without the use of laxatives for ≥ 6 months prior to preliminary enrollment
* Patients who underwent pancolonoscopy or contrast enema after development of the CC symptoms and within 5 years prior to preliminary enrollment, and in whom no organic change was observed which dose not influence on CC symptoms
* Female patients must be either:

If of non-childbearing potential:

* Post-menopausal at the preliminary enrollment, or documented surgically sterile Or, if of childbearing potential,
* Agree not to try to become pregnant during the study and for 28 days after the final study drug administration
* And have a negative urine pregnancy test at screening
* And, if heterosexually active, agree to consistently use two forms of highly effective birth control throughout the study period and for 28 days after the final study drug administration

  * Female patients must agree not to breastfeed throughout the study period and for 28 days after the final study drug administration
  * Female patients must not donate ova starting throughout the study period and for 28 days after the final study drug administration
  * Male subject and their female spouse/partners who are of childbearing potential must be using two forms of highly effective form of birth control starting at Screening and continue throughout the study period, and for 28 days after the final study drug administration
  * Male subject must not donate sperm starting at Screening and throughout the study period and, for 28 days after the final study drug administration

Exclusion Criteria:

* Patients who have met the Rome III diagnostic criteria for IBS; with recurrent abdominal pain or discomfort for ≥ 3 days/month in the last 3 months prior to preliminary enrollment, associated with ≥ 2 of the 3 characteristics described below and with the symptoms (IBS symptoms) described above for ≥ 6 months prior to preliminary enrollment

  1. Improvement with defecation
  2. Onset associated with a change in frequency of stool
  3. Onset associated with a change in form (appearance) of stool
* Patients with a history of surgical resection of the stomach, gallbladder, small intestine, or large intestine
* Patients with a history or current evidence of inflammatory bowel disease or ischemic colitis
* Patients with concurrent infectious enteritis, hyperthyroidism or hypothyroidism, constipation due to anorectal dysfunction, drug-induced constipation, constipation due to other organic diseases or active peptic ulcer
* Patients with apparent mechanical obstruction
* Patients with megacolon or megarectum
* For female patients, patients with concurrent endometriosis or adenomyosis
* Patients who are considered to have severe depression or a severe anxiety disorder that can affect the efficacy evaluation of the study drug
* Patients with a history of abuse of drugs or alcohol, or current abuse of drugs or alcohol
* Patients who used/underwent or are scheduled to use/undergo prohibited concomitant drugs or therapies, or in whom prohibited examinations were conducted or are scheduled to be conducted 3 days prior to the start of the bowel habit observation period
* Patients with a history or current evidence of malignant tumors
* Patients with concurrent serious cardiovascular diseases, respiratory diseases, renal diseases, hepatic diseases, gastrointestinal disorders, blood diseases, or neurological/psychiatric diseases
* Patients with a history of drug allergies
* Patients who have participated in the clinical trial of ASP0456 or have been administered ASP0456
* Patients who have participated or are participating in another clinical trial or post-marketing clinical study of other ethical drugs or medical devices within 12 weeks prior to obtaining informed consent

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2016-06-24 (Actual); Primary Completion 2016-11-14 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in weekly mean SBM frequency during one week of administration (Part I) | Baseline and Week 1
  SBM: Spontaneous bowel movement

SECONDARY OUTCOMES:
Change from baseline in weekly mean SBM frequency | Baseline and up to Week 56
Weekly responder rate of SBM | Baseline and up to Week 56
  The weekly average value of SBM frequency is more than 3 and over 1 more than the weekly mean value of SBM frequency in the bowel habit observation period.
Percentage of subjects with SBM within 24 hours after the start of the initial administration | Up to 24h
Time to first SBM | Up to Week 4
Change from baseline in weekly mean CSBM frequency | Baseline and up to Week 56
  CSBM: SBM without a sensation of incomplete evacuation
Weekly responder rate of CSBM | Baseline and up to Week 56
  The weekly average value of CSBM frequency is more than 3 and over 1 more than the weekly mean value of CSBM frequency in the bowel habit observation period.
Percentage of subjects with CSBM within 24 hours after the start of the initial administration | Up to 24h
Change from baseline in weekly mean stool form score | Baseline and up to Week 56
  Stool form will be measured using seven-point Bristol Stool Form Scale.
Change from baseline in weekly mean abdominal bloating severity score | Baseline and up to Week 56
  Abdominal bloating severity will be measured using a five-point ordinal score.
Change from baseline in weekly mean abdominal pain/discomfort severity score | Baseline and up to Week 56
  Abdominal pain/discomfort severity will be measured using a five-point ordinal score.
Change from baseline in weekly mean straining severity score | Baseline and up to Week 56
  Straining severity will be measured using a five-point ordinal score.
Weekly responder rate of global assessment of relief of CC symptoms | Up to Week 56
  CC: chronic constipation; The weekly responder of the evaluation items shall be the subject satisfying the following at the time of evaluation in each week: Score of Global assessment of relief of chronic constipation symptoms (7 scores: 1-7) is 1 or 2.
Weekly responder rate of abnormal bowel habits improvement in CC | Up to Week 56
  Score of abdominal bowel habits improvement effect (7 scores: 1-7) is 1 or 2.
Weekly responder rate of abdominal symptoms relief of CC | Up to Week 56
  Score of abdominal symptom improvement effect (7 scores: 1-7) is 1 or 2.
Change from baseline in IBS-QOL-J score | Baseline and up to Week 56
  IBS-QOL-J: Japanese version of Irritable Bowel Syndrome Quality of Life
Safety assessed by incidence of adverse events | Up to Week 56
Number of participants with abnormal Vital signs and/or adverse events during treatment period | Up to Week 56
Number of participants with abnormal Laboratory values and/or adverse events during treatment period | Up to Week 56
Safety assessed by body weight | Up to Week 56

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (39):
- Japan (39):
  - Site JP00029, Aichi
  - Site JP00030, Aichi
  - Site JP00021, Chiba
  - Site JP00022, Chiba
  - Site JP00023, Chiba
  - Site JP00024, Chiba
  - Site JP00040, Fukuoka
  - Site JP00001, Hokkaido
  - Site JP00002, Hokkaido
  - Site JP00037, Hyōgo
  - Site JP00038, Hyōgo
  - Site JP00039, Hyōgo
  - Site JP00017, Kanagawa
  - Site JP00018, Kanagawa
  - Site JP00019, Kanagawa
  - Site JP00020, Kanagawa
  - Site JP00031, Osaka
  - Site JP00032, Osaka
  - Site JP00033, Osaka
  - Site JP00034, Osaka
  - Site JP00035, Osaka
  - Site JP00036, Osaka
  - Site JP00025, Saitama
  - Site JP00026, Saitama
  - Site JP00027, Saitama
  - Site JP00028, Saitama
  - Site JP00003, Tokyo
  - Site JP00004, Tokyo
  - Site JP00005, Tokyo
  - Site JP00006, Tokyo
  - Site JP00007, Tokyo
  - Site JP00008, Tokyo
  - Site JP00009, Tokyo
  - Site JP00010, Tokyo
  - Site JP00011, Tokyo
  - Site JP00012, Tokyo
  - Site JP00013, Tokyo
  - Site JP00014, Tokyo
  - Site JP00015, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=280